CLINICAL TRIAL: NCT04799652
Title: Are Surgeons Ready to Get the COVID-19 Vaccine?
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Pierre Wauthy, Medical Director of the CHU Brugmann, Brugmann University Hospital
Other Study IDs: CHUB-Farid-vaccination
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Doctors within Belgian Hospitals
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey of 21 questions. The questions were divided into sections, evaluating demographics, COVID-19 test status and symptoms, the surgeon's opinion on the COVID-19 vaccination and their main concerns. The questionnaire was completed anonymously between 15/01/2021 and 24/01/2021, before the start of vaccination of health care professionals in a Belgian hospital.

SUMMARY:
The COVID-19 pandemic continues to rage and most of the world is facing a second wave with continuous lockdown and strict measures aiming to control it. While vaccination is on its way, and has even started in several countries, trust and acceptance remain a challenge for an effective vaccination strategy, especially with the increasing vaccination hesitance in recent years . It is important to understand the main concerns towards the COVID-19 vaccine so they can be addressed in a constructive way - more specifically among health care professionals who are at the frontline of the pandemic.

The aim of this study is to evaluate whether surgeons are ready for the COVID-19 vaccine and to understand their main concerns towards the vaccine.

In an objective to evaluate the attitude of doctors towards the COVID vaccine and the effect of prolonged lockdown on their psychological burden, the investigators created an anonymous survey of 21 questions.

ELIGIBILITY:
Inclusion Criteria:

* Physicians affiliated to Belgian Hospitals

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians affiliated to Belgian Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Perception and knowledge towards the vaccine | 15 minutes
  Survey (21 items). Qualitative questionnaire about the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Farid, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No